CLINICAL TRIAL: NCT01382849
Title: F-18-AV-45 Uptake, Spot Sign Presence and Cerebral Amyloid Angiopathy (CAA) in Primary Intracranial Hemorrhage (ICH)
Status: Withdrawn | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Richard I Aviv, Sunnybrook Hospital
Other Study IDs: 18F-AV-45-A14
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Cerebral Amyloid Angiopathy
Keywords: amyloid; cerebral amyloid angiopathy; hemorrhages; cerebral spot sign
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Alzheimer Disease; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CAA positive microbleeders: Cerebral amyloid angiopathy (CAA) positive microbleeders
- probable CAA macrobleeders
- CAA negative microbleeders

SUMMARY:
Florbetapir F 18 is an experimental radioactive drug that may allow doctors to image changes in the brain using a PET (Positron Emission Tomography) scanner. The purpose of this study is to evaluate the imaging characteristics of, Florbetapir F 18 (also known as 18F-AV-45) in patients who have previously undergone bleeding in their brains. Florbetapir F 18 binds to amyloid-ß peptide (Aß) that accumulates in the brains of patients with bleeding. These accumulations are called amyloid plaques and when extensive are labeled cerebral amyloid angiopathy (CAA). Florbetapir F 18 sticks to the amyloid plaques in the brain and emits a low level of gamma rays which can be detected by a PET camera.

MRI detected microbleeds have been identified as markers of clinically silent hemorrhage from bleeding-prone vessels. Another imaging marker of vessel damage and risk of bleeding is the spot sign (SS). Finally, certain genetic signatures (ApoE genotype) have been shown to be associated with Aß deposition in the brain or predispose patients to higher risks of bleeding. This research study will explore the interactions of these factors and understand the physiology of intracerebral bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Prior intracranial hemorrhage at least 3 months prior
* Patients >18 years

Exclusion Criteria:

1. Modified Rankin score >3.
2. Clinically significant medical comorbidities which in the opinion of the investigator might pose a potential safety risk to the subject.
3. Women of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception.
4. Have a history of relevant severe drug allergy or hypersensitivity
5. Patients who withdraw consent. Age and gender-matched microbleed patients previously demonstrating MRI microbleeds without prior macrobleeds will be recruited from stroke clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Macrobleed patients will be selected from a prospectively maintained ICH database at Sunnybrook Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Type of Bleed | 2-3 weeks
  Patients will be divided into micro- and macro- bleeders based on MRI detected microhemorhage pattern. Processing of each patient will take 2-3 weeks.
Spot Sign Status | 2-3 weeks
  They will be further subdivided by spot sign status into positive or negative.
Amyloid uptake | 2-3 weeks

SECONDARY OUTCOMES:
ApoE genotype | 2-3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aviv, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada